CLINICAL TRIAL: NCT00339872
Title: Randomized, Double-Blind, Placebo-Controlled, Sequential-Group, Ascending Single Dose Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IMA-638 Administered Subcutaneously and Intravenously to Subjects With Asthma
Brief Title: Study Evaluating IMA-638 in Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: 3174K1-100
Record Dates: First submitted 2006-06-20; First posted 2006-06-21 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-12

CONDITIONS: Asthma
Keywords: healthy subjects
MeSH Terms: conditions — Asthma | interventions — anrukinzumab

INTERVENTIONS:
Drug: IMA-638

SUMMARY:
The purpose of this study is to evaluate the safety of, and blood drug levels for, single, ascending doses of IMA-638 in mild to moderate asthma subjects.

ELIGIBILITY:
Inclusion Criteria:

* Men and women of non-childbearing potential with mild to moderate asthma as defined by forced expiratory volume in 1 second (FEV1) greater than 70% predicted.
* Well controlled asthma, as exhibited by completion of asthma questionnaire.
* Otherwise healthy, except for asthma.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2006-02; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Safety will be measured by evaluating physical examinations, spirometry, vital signs, electrocardiograms (ECGs), and clinical laboratory test results.

SECONDARY OUTCOMES:
Drug levels in the blood and associated biomarkers will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Denver, Colorado, United States